CLINICAL TRIAL: NCT04104282
Title: the Role of plin5 in the Development of a Sequence Polymorphism in Patatin-like Phospholipid Domain Containing Protein 3 Polymorphism-associated Nonalcoholic Fatty Liver Disease
Brief Title: the Role of plin5 in the Development of Nonalcoholic Fatty Liver Disease.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY-20162068-2
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2019-07

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Nonalcoholic fatty liver disease; Lipid droplets; Plin5
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To further clarify the role of sequence polymorphism in patatin-like phospholipid domain containing protein 3 in the development of nonalcoholic fatty liver disease.

DETAILED DESCRIPTION:
A sequence polymorphism in patatin-like phospholipid domain containing protein 3 is significantly associated with nonalcoholic fatty liver disease, but its mechanism underlying this association remains obscure. We introduce the human samples of liver to clarify the relationship between the expression of plin5 and the development of sequence polymorphism in patatin-like phospholipid domain containing protein 3 variant-associated nonalcoholic fatty liver disease, analyze the lipid metabolism and lipotoxicity of hepatocytes to elucidate the mechanisms of plin5 in the development of sequence polymorphism in patatin-like phospholipid domain containing protein 3 variant-associated nonalcoholic fatty liver disease. Our study will contribute to the mechanism of nonalcoholic fatty liver disease, and its prevention and therapy.

ELIGIBILITY:
Inclusion criteria:

The diagnosis of simple fatty liver disease was confirmed by clinical presentation, ultrasound, and without long-term drinking history, viral hepatitis, medication history, obesity (BMI≥30), type 2 diabetes and other metabolic diseases.

Exclusion criteria:

With long-term drinking history, viral hepatitis, medication history, obesity (BMI≥30), type 2 diabetes and other metabolic diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with was confirmed by clinical presentation, ultrasound and laboratory test. At the same time, participants who enrolled this statistical analysis without long-term drinking history, viral hepatitis, medication history, obesity (BMI≥30), type 2 diabetes and other metabolic diseases. (range, 18-75 years).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2025-12-27 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
The severity of non-alcoholic fatty liver disease | 3 months
  Evaluating by ultrasound the severity of non-alcoholic fatty liver disease

SECONDARY OUTCOMES:
The expression of plin5 | 3 months
  Evaluating by biochemical methods the expression of plin5 in patients liver tissue

CONTACTS AND LOCATIONS:
Overall Officials: Ming Yu, PhD, MD, Study Director — The Xijing Hospital of Fourth Military Medical University
Locations (1):
- The Department of Ultrasonic Medicine, The Xijing Hospital of Fourth Military Medical University, Xi'an, Shaanxi, China